CLINICAL TRIAL: NCT06970990
Title: Use of Nasal Pressure to Assess Inspiratory Effort Under Different Oxygen Treatments: a Prospective Physiological Study
Brief Title: Use of Nasal Pressure to Assess Inspiratory Effort Under Different Oxygen Treatments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jian-Xin Zhou (Other)
Responsible Party: Sponsor-Investigator, Jian-Xin Zhou, Head of Emergency and Critical Care Center, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IIT2025-031-002
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Critical Care; Inspiratory Effort
Keywords: Esophageal pressure; inspiratory effort; oxygen treatments; Nasal Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- HFNC:flow=50L/min (Experimental): Under high-flow oxygen therapy at a flow rate of 50 L/min, record/monitor for 5 minutes
  Interventions: Procedure: HFNC:50L/min
- HFNC:flow=40L/min (Experimental): Under high-flow oxygen therapy at a flow rate of 40 L/min, record/monitor for 5 minutes
  Interventions: Procedure: HFNC:flow=40L/min
- HFNC:flow=30L/min (Experimental): Under high-flow oxygen therapy at a flow rate of 30 L/min, record/monitor for 5 minutes
  Interventions: Procedure: HFNC:flow=30L/min
- Face Mask Oxygen:8L/min (Experimental): Under face mask oxygen at a flow rate of 8 L/min, record/monitor for 5 minutes.
  Interventions: Procedure: Face mask oxygen:8L/min
- Face Mask Oxygen:5L/min (Experimental): Under face mask oxygen at a flow rate of 5 L/min, record/monitor for 5 minutes.
  Interventions: Procedure: Face mask oxygen:5L/min
- Nasal cannula oxygen:5L/min (Experimental): Under nasal cannula oxygen at a flow rate of 5 L/min, record/monitor for 5 minutes.
  Interventions: Procedure: Nasal cannula oxygen:5L/min
- Nasal cannula oxygen:3L/min (Experimental): Under nasal cannula oxygen at a flow rate of 3 L/min, record/monitor for 5 minutes.
  Interventions: Procedure: Nasal cannula oxygen:3L/min

INTERVENTIONS:
Procedure: HFNC:50L/min — Under high-flow oxygen therapy at a flow rate of 50 L/min, record/monitor for 5 minutes
  Arms: HFNC:flow=50L/min
Procedure: HFNC:flow=40L/min — Under high-flow oxygen therapy at a flow rate of 40 L/min, record/monitor for 5 minutes.
  Arms: HFNC:flow=40L/min
Procedure: HFNC:flow=30L/min — Under high-flow oxygen therapy at a flow rate of 30 L/min, record/monitor for 5 minutes.
  Arms: HFNC:flow=30L/min
Procedure: Face mask oxygen:8L/min — Under face mask oxygen at a flow rate of 8 L/min, record/monitor for 5 minutes.
  Arms: Face Mask Oxygen:8L/min
Procedure: Face mask oxygen:5L/min — Under face mask oxygen at a flow rate of 5 L/min, record/monitor for 5 minutes.
  Arms: Face Mask Oxygen:5L/min
Procedure: Nasal cannula oxygen:5L/min — Under nasal cannula oxygen at a flow rate of 5 L/min, record/monitor for 5 minutes.
  Arms: Nasal cannula oxygen:5L/min
Procedure: Nasal cannula oxygen:3L/min — Under nasal cannula oxygen at a flow rate of 3 L/min, record/monitor for 5 minutes.
  Arms: Nasal cannula oxygen:3L/min

SUMMARY:
The aim of this study was to investigate the effects of different oxygen therapy modalities (including nasal cannula oxygen, mask oxygen and high-flow nasal cannula oxygen) on the correlation between Nasal Pressure and Esophageal Pressure by means of a prospective physiological study, to assess the dynamic changes of nasal pressure and esophageal pressure and their underlying mechanisms under different conditions of oxygen therapy, to analyse the effects of oxygen therapy parameters on the relationship between the two, and to explore the feasibility of nasal pressure as a non-invasive monitoring indicator, in order to replaceor supplement esophageal manometry in clinical practice, especially in patients with respiratory distress and instability.Meanwhile, this study will also evaluate the effects of different oxygen therapy modalities on patients' respiratory mechanics and comfort, provide a scientific basis for the clinical selection of individualised oxygen therapy regimens, and ultimately provide new physiological evidence for the management of oxygen therapy in patients with acute respiratory failure in the intensive care unit (ICU) and outside the ICU, promote the development of non-invasive monitoring technology, and improve the clinical prognosis and therapeutic experience of patients.

DETAILED DESCRIPTION:
Patients in the intensive care unit (ICU) often require different modalities of oxygen therapy to maintain adequate oxygenation.Common oxygen therapy modalities include nasal cannula oxygen, face mask oxygen and high flow nasal cannula oxygen (HFNC).These modalities of oxygen therapy not only affect the patient's oxygenation status, but may also influence nasal and esophageal pressures by altering the upper airway pressure gradient, which in turn affects respiratory mechanics and patient comfort.

Esophageal pressure fluctuations (ΔPes), as a reflection of mean transpulmonary pressure during unassisted voluntary breathing, provide an important basis for assessing inspiratory effort.However, esophageal manometry still faces many challenges for its bedside implementation in clinical practice, especially in unstable patients with respiratory distress and severely impaired gas exchange.Notably, the COVID-19 pandemic has led to a significant increase in the number of patients with acute respiratory failure, who often require condition-specific oxygen therapy of varying severity and are mostly treated outside the ICU.Given that such patients are at high risk of deterioration, it is particularly important to continuously monitor their inspiratory effort.

nasal pressure is an important physiological indicator for assessing upper airway resistance and airflow dynamics characteristics, whereas esophageal pressure is a key parameter that directly reflects intrathoracic pressure and respiratory effort.Previous studies have shown that there may be a physiological correlation between intranasal pressure and oesophageal pressure, and that this correlation may be influenced by a variety of factors, including airflow velocity, oxygen concentration, and the dynamics of upper airway resistance.Earlier physiological studies by comparing oesophageal pressure fluctuations (ΔPes) with nasal pressure fluctuations (ΔPnose) fluctuations found that when inspiratory effort was increased, there was no significant phase difference between these pressure waveforms.In addition, it was observed that there was a significant correlation between ΔPes and airway pressure fluctuations (ΔPaw) obtained by airway occlusion manoeuvres during inspiratory effort testing.However, although these findings provide important clues for understanding respiratory mechanics, studies on the correlation between nasal pressure and esophageal pressure under different oxygen therapy conditions are still relatively limited, especially lacking data support from prospective physiological studies.Therefore, further systematic studies are needed in the future to investigate in depth the effects of different oxygen therapy parameters (e.g., flow rate, humidity, and temperature, etc.) on the relationship between nasal pressure and esophageal pressure, so as to provide more precise guidance for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. No mechanical ventilation required,Able to tolerate oxygen therapy via nasal cannula, standard face mask, or nasal high-flow oxygen therapy;
2. Respiratory stability:Capable of spontaneous breathing with effective cough for secretion clearance.Oxygen saturation (SpO₂) > 90% or PaO₂/FiO₂ ≥ 150 mmHg when receiving nasal cannula oxygen at 3 L/min;
3. Hemodynamic stability:Heart rate (HR) ≤ 120 bpm;Systolic blood pressure (SBP) 90-150 mmHg;No vasoactive medications OR norepinephrine dosage < 0.1-0.2 μg/kg·min (or equivalent doses of other vasoactive agents);
4. Metabolic stability;
5. Compliance with medical instructions.Able to follow prescribed tasks.Esophageal pressure monitoring catheter already in place;
6. Patient or legal guardian agrees to participate and has signed the informed consent form.

Exclusion Criteria:

1. Age < 18 years;
2. Pregnancy;
3. Hemodynamic instability:Mean arterial pressure (MAP) < 60 mmHg.Heart rate (HR) > 120 bpm or < 60 bpm;
4. Respiratory instability:Respiratory rate (RR) > 35 bpm.Oxygen saturation (SpO₂) < 90%;
5. Neuromuscular diseases or phrenic nerve injury;
6. Recent trauma or surgery involving the trachea, esophagus, neck, or chest.Contraindications to esophageal catheter placement or inability to monitor esophageal pressure;
7. Nasal obstruction or anatomical abnormalities:Complete nasal obstruction.Severe anatomical abnormalities (e.g., severe septal deviation, nasal polyps, or tumors) preventing catheter placement or compromising ventilation;
8. High-risk craniofacial conditions:Severe facial trauma or skull base fracture with risk of catheter misplacement into the intracranial space.Active epistaxis or incomplete healing after nasal surgery;
9. Bleeding risk:Severe coagulopathy.Esophageal/gastric varices or other conditions predisposing to hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tidal swing of nasal cuff pressure (ΔPnose) | From enrollment to the end of treatment at 4 hours
  Tidal swing of nasal pressure (ΔPnose) will be measured
Tidal swing of esophageal pressure (∆Pes) | From enrollment to the end of treatment at 4 hours
  Tidal swing of esophageal pressure (∆Pes) will be measured

SECONDARY OUTCOMES:
Respiratory rate | From enrollment to the end of treatment at 4 hours.
  Respiratory rate will be measured at each type of oxygen treatment.
COMFORT scale | From enrollment to the end of treatment at 4 hours
  COMFORT scale will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No